CLINICAL TRIAL: NCT05666258
Title: Gene Expression Profiling to Help Define the Need for Neo-Adjuvant Chemotherapy in HR+, HER- Breast Cancer Patients
Acronym: NACAGEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: NACAGEP
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy; GEP
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: GEP — GEP before surgery to determine need for neoadjuvant chemotherapy
  Other Names: Mammaprint

SUMMARY:
The goal of the experiment is surgical de-escalation. Patients with newly diagnosed cT1-3, cN1, cM0 and HR+, HER2- breast cancer and low clinical risk usually first receive breast cancer surgery, after which chemotherapy can be added based on the final anatomopathological results or additional Gene Expression Profiling (GEP) testing.

Chemotherapy helps reduce the cancer recurrence or metastasis risk. Adjuvant chemotherapy (AC) can be given for large tumours, aggressive tumours with high grade tumour cells, or if axillary lymph node invasion is discovered during surgery. If the investigators were able to identify patients requiring chemotherapy prior to surgery, they could treat them with Neo-Adjuvant Chemotherapy (NAC) instead. By using MammaPrint® GEP, the investigators would be able to stratify patients into either a low- or high-risk category. Since the high-risk group is known to benefit from chemotherapy to improve overall survival, they would be treated with NAC, which could also potentially lead to surgical de-escalation. Breast conserving procedures, such as a lumpectomy instead of a mastectomy, could allow more aesthetically pleasing results and increase patient quality of life. Using NAC for patients with axillary lymph node invasion could lead to nodal complete pathological response (cN1 -> ypN0), allowing patients that are willing to enter the TADANAC trial a lymph node sparing procedure instead of a full axillary lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Tumour characteristics: HR+, HER-
* Histopathological tumour characteristics: cT1-3, cN1, cM0, all histological types included
* Age: 18-85 years

Exclusion Criteria:

* Tumour characteristics: cT4, cN2-3, cM1
* Age: <18 or >85 years old
* Received chemotherapy in the last 5 years
* Pregnancy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Breast Clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-11-14 (Estimated); Study Completion 2024-11-14 (Estimated)

PRIMARY OUTCOMES:
De-escalation of breast cancer surgery | 8 months after inclusion
  Number of patients who receive NAC after a high-risk GEP that will undergo TAD instead of ALND and/or undergo BCS instead of mastectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium